CLINICAL TRIAL: NCT02974569
Title: Improving Symptom Self-management in Adolescents & Young Adults With Cancer
Acronym: CSCAT2
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); St. Baldrick's Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: MCC-16-12876; HM20007402 (Other: IRB)
Record Dates: First submitted 2016-11-06; First posted 2016-11-28 (Estimated); Last update posted 2017-12-22 (Actual); Status verified 2017-12

CONDITIONS: Symptom Clusters; Cancer
Keywords: adolescents; young adults
MeSH Terms: conditions — Syndrome; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- C-SCAT: C-SCAT arm: Completes and uses Computerized Symptom Capture Tool (C-SCAT) during visit with provider for two clinic visits.
  Interventions: Device: Computer Symptom Capture Tool

INTERVENTIONS:
Device: Computer Symptom Capture Tool — C-SCAT is an investigator developed app that is delivered via an iPad. The original CSCAT included the 30 symptoms from the Memorial Symptom Assessment Scale. The recently updated version includes two additional symptoms "feeling bloated" and "sexual dysfunction" that are included in the adult version of the MSAS.21 These symptoms were added based on feedback from the initial AYA sample of 13-29 year olds and in consideration of the developmental perspectives of the AYA population.The CSCAT allows the user to create an image of his or her symptom experience.
  Other Names: C-SCAT

SUMMARY:
This study evaluates the use of the Computerized Symptom Capture Tool (C-SCAT), which creates an image of the symptoms the participant is experiencing, for improving symptom self-management in adolescents and young adults with cancer. In this one-group trial, participants will complete the C-SCAT and use it during two clinic visits with their oncology providers.

DETAILED DESCRIPTION:
Unrelieved symptoms lead to poorer quality of life for adolescents and young adults (AYAs) with cancer. Strategies are needed to help AYAs manage symptoms. The investigators developed the Computerized Symptom Capture Tool (C-SCAT), a novel way to assess symptoms where AYAs create a picture of their symptoms using images and text on an iPad app. The resulting image shows symptoms/symptom clusters, priority symptoms and relationships between symptoms and has potential to support AYA's symptom self-management. Facilitating the self-management process, including self-efficacy, self-regulation behaviors, and patient-provider communication, is essential for improving symptom outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 15 to 29 years of age with a diagnosis of cancer (primary, relapsed/recurrent, refractory, progressive, or secondary malignancy) receiving myelosuppressive chemotherapy.
* Completion of at least one cycle of therapy for cancer and anticipated to have at least two additional cycles of myelosuppressive chemotherapy as part of the treatment plan.
* Ability to speak and understand English as required to complete the C-SCAT and study measures.
* Ability to use a tablet computer.

Exclusion Criteria:

* Cognitive and/or physical inabilities to complete the proposed study measures as determined by self--report, parent report of minor, or medical chart.

Ages: 15 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric and adult oncology clinics at the Virginia Commonwealth University Health System (VCUHS). Patients and parents of minor patients will be approached as inpatients or as outpatients at Massey Cancer Center Fellows Clinic and at the Pediatric Oncology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-10-25 (Actual); Study Completion 2017-10-25 (Actual)

PRIMARY OUTCOMES:
Change in self-efficacy of symptom management measured by PROMIS Self-efficacy of symptom management scale. | Baseline, immediately after first provider visit (approx. 2 -4 weeks from baseline) and then immediately after second provider visit (approx. 6-8 weeks from baseline)
Change in patient-provider communication from patient perspective measured by Patient-Provider Communication Scale. | Baseline, immediately after first provider visit (approx. 2 -4 weeks from baseline) and then immediately after second provider visit (approx. 6-8 weeks from baseline)
Change in self-regulation of symptoms assessed by an audio-taped semi-structured interview. | Within 24 hours after first provider visit (approx. 2 -4 weeks from baseline) and Within 24 hours after second provider visit (approx. 6-8 weeks from baseline)
  Semi-structured interviews to address how using the C-SCAT impacts self-regulation behaviors, such as self-monitoring, reflective thinking, and decision-making
Change in provider's usefulness of using C-SCAT assessed by Provider Questionnaire. | After first provider visit (approx. 2 -4 weeks from baseline) and after second provider visit (approx. 6-8 weeks from baseline)
Change in provider's usefulness of using C-SCAT assessed by providers' documentation of symptoms in the electronic health record. | After first provider visit (approx. 2 -4 weeks from baseline) and after second provider visit (approx. 6-8 weeks from baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne W. Ameringer, Ph.D., Principal Investigator — Virginia Commonwealth University
Locations (2):
- United States (2):
  - The Childrens Mercy Hospital, Kansas City, Missouri
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia